CLINICAL TRIAL: NCT05500352
Title: Myocardial Work and Left Ventricular Mechanical Dyssynchrony During Acute Changes in Plasma Glucose in Individuals With Type 1 Diabetes, Type 2 Diabetes and Without Diabetes
Brief Title: Acute Changes in Plasma Glucose and Cardiovascular Disease in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H18034040_part2
Record Dates: First submitted 2022-07-06; First posted 2022-08-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Diabetes; Hypoglycemia; Hyperglycemia; Cardiovascular Diseases; Sudden Cardiac Death
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Hyperglycemia; Cardiovascular Diseases; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: The present echocardiographic study includes participants from three experimental clamp studies; the Hypo-Heart 1 (Study 1), Hypo-Heart 2 (Study 2) and Rapid-Heart (Study 3).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cardiovascular effects of slowly declining plasma glucose in type 1 diabetes (Experimental)
  Interventions: Other: Hyperglycemia with slow decline in plasma glucose in type 1 diabetes
- Cardiovascular effects of rapidly declining plasma glucose in type 1 diabetes (Experimental)
  Interventions: Other: Hyperglycemia with rapid decline in plasma glucose in type 1 diabetes
- Cardiovascular effects of rebound hyperglycemia in type 1 diabetes (Experimental)
  Interventions: Other: Rebound hyperglycemia in type 1 diabetes
- Cardiovascular effects of rebound euglycemia in type 1 diabetes (Experimental)
  Interventions: Other: Rebound euglycemia in type 1 diabetes
- Cardiovascular effects of hypoglycemia in type 1 diabetes (Experimental)
  Interventions: Other: Hypoglycemia in type 1 diabetes
- Cardiovascular effects of hypoglycemia in type 2 diabetes (Experimental)
  Interventions: Other: Hypoglycemia in type 2 diabetes
- Cardiovascular effects of hypoglycemia in healthy controls (Experimental)
  Interventions: Other: Hypoglycemia in healthy controls
- Cardiovascular effects of hyperglycemia in type 2 diabetes (Experimental)
  Interventions: Other: Hyperglycemia in type 2 diabetes
- Cardiovascular effects of hyperglycemia in healthy controls (Experimental)
  Interventions: Other: Hyperglycemia in healthy controls

INTERVENTIONS:
Other: Hyperglycemia with slow decline in plasma glucose in type 1 diabetes — Acute plasma glucose decline, divided into the following three phases: 1) Hyperglycaemic phase (plasma glucose 15 mmol/l), 2) Slow plasma glucose decline phase and 3) Euglycaemic phase (plasma glucose 4.5-5.5 mmol/l).
  Arms: Cardiovascular effects of slowly declining plasma glucose in type 1 diabetes
Other: Hyperglycemia with rapid decline in plasma glucose in type 1 diabetes — Acute plasma glucose decline, divided into the following three phases: 1) Hyperglycaemic phase (plasma glucose 15 mmol/l), 2) Rapid plasma glucose decline phase and 3) Euglycaemic phase (plasma glucose 4.5-5.5 mmol/l).
  Arms: Cardiovascular effects of rapidly declining plasma glucose in type 1 diabetes
Other: Rebound hyperglycemia in type 1 diabetes — Includes three steady state phases in plasma glucose, 1) euglycemic phase (5-8 mmol/L), 2) hyperinsulinemic hypoglycemic phase (PG: 2.5 mmol/L), 3) recovery phase in hyperglycemia (20.0 mmol/L)
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of rebound hyperglycemia in type 1 diabetes
Other: Rebound euglycemia in type 1 diabetes — Includes three steady state phases in plasma glucose, 1) euglycemic phase (5-8 mmol/L), 2) hyperinsulinemic hypoglycemic phase (PG: 2.5 mmol/L), 3) recovery phase in euglycemia (PG: 5-8 mmol/L).
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of rebound euglycemia in type 1 diabetes
Other: Hypoglycemia in type 1 diabetes — Includes three steady state phases in plasma glucose, 1) euglycemic phase (5-8 mmol/L), 2) hyperinsulinemic hypoglycemic phase (PG: 2.5 mmol/L), 3) recovery phase in hyperglycemia (20.0 mmol/L) or euglycemia (PG: 5-8 mmol/L)
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of hypoglycemia in type 1 diabetes
Other: Hypoglycemia in type 2 diabetes — Includes three steady state phases in plasma glucose, 1) euglycemic phase (fasting PG), 2) hyperglycemic phase (fasting PG + 10 mmol/L), 3) hyperinsulinemic hypoglycemic phase (PG < 3.0 mmol/L).
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of hypoglycemia in type 2 diabetes
Other: Hypoglycemia in healthy controls — Includes three steady state phases in plasma glucose, 1) euglycemic phase (fasting PG), 2) hyperglycemic phase (fasting PG + 10 mmol/L), 3) hyperinsulinemic hypoglycemic phase (PG < 3.0 mmol/L).
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of hypoglycemia in healthy controls
Other: Hyperglycemia in type 2 diabetes — Includes three steady state phases in plasma glucose, 1) euglycemic phase (fasting PG), 2) hyperglycemic phase (fasting PG + 10 mmol/L), 3) hyperinsulinemic hypoglycemic phase (PG < 3.0 mmol/L).
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of hyperglycemia in type 2 diabetes
Other: Hyperglycemia in healthy controls — Includes three steady state phases in plasma glucose, 1) euglycemic phase (fasting PG), 2) hyperglycemic phase (fasting PG + 10 mmol/L), 3) hyperinsulinemic hypoglycemic phase (PG < 3.0 mmol/L).
  Other Names: Experimental clamp
  Arms: Cardiovascular effects of hyperglycemia in healthy controls

SUMMARY:
Patients with diabetes have an increased risk of sudden cardiac death compared to the general population. Severe hypoglycemia is associated with an increased risk of cardiovascular (CV) disease (CVD) and events, including cardiac arrhythmias and sudden cardiac death; likewise, increased glycemic variability is associated with macrovascular complications and increased mortality. The physiological mechanisms linking hypoglycemia and glycemic variability to CVD and CV events remain unclear.

Myocardial work and mechanical dyssynchrony will be measured by speckle tracking echocardiography during euglycemia, hypoglycemia and hyperglycemia in individuals with type 1 diabetes, type 2 diabetes, and without diabetes. Echocardiographic images from three experimental clamp studies - Hypo-Heart 1 (sub-study 1), Hypo-Heart 2 (sub-study 2) and Rapid-Heart - will be included in this study.

DETAILED DESCRIPTION:
The results of this study may be compiled into one or more manuscripts for publication.

Study ID's:

Hypo-Heart 1 (sub-study 1): NCT03956173 Hypo-Heart 2 (sub-study 2): NCT03150030 Rapid-Heart: NCT04800536

ELIGIBILITY:
The present echocardiographic study includes 86 participants from three experimental clamp studies; the Hypo-Heart 1 (Study 1), Hypo-Heart 2 (Study 2) and Rapid-Heart (Study 3), including patients with type 1 diabetes (Hypo-Heart 1 and Rapid-Heart), patients with type 2 diabetes (Hypo-Heart 2) and healthy controls (Hypo-Heart 2).

Hypo-Heart 1:

Inclusion Criteria:

* Informed and written consent
* Type 1 diabetes diagnosed according to the criteria of the World Health Organization (WHO)
* Age 18-70 years
* Insulin treatment for ≥3 years

Exclusion Criteria:

* Arrhythmia diagnosed prior to the screening visit
* Implantable cardioverter defibrillator (ICD) or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated eltroxin substituted myxoedema)
* Anemia (male: hemoglobin <8.0; female: hemoglobin <7.0 mmol/l)

Hypo-Heart 2:

Inclusion Criteria: Patients with type 2 diabetes

* Informed and written consent
* Type 2 diabetes diagnosed according to the criteria of the World Health Organization (WHO)
* Treatment with insulin
* Glycated haemoglobin A1c (HbA1c) ≤58 mmol/mol

Inclusion Criteria: Healthy individuals

* HbA1c ≤42 mmol/mol
* Fasting plasma glucose ≤6.1 mmol/l

Exclusion Criteria: Patients with type 2 diabetes

* Arrhythmia diagnosed prior to or at the time of inclusion
* Implantable cardioverter defibrillator (ICD) or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Insulin naïve patients with type 2 diabetes
* Thyroid dysfunction (except for well-regulated eltroxine substituted myxoedema)
* Unable to comply with daily CGM during run-in period
* Anemia (male: hemoglobin < 8.0; female: hemoglobin < 7.0 mmol/l)

Exclusion Criteria: Healthy individuals

* Type 1 or type 2 diabetes
* Prediabetes (HbA1c >42 mmol/l and/or fasting plasma glucose >6.1 mmol/l)
* Family history of diabetes (type 1 og type 2 diabetes)
* Arrhythmia diagnosed prior to or at the time of inclusion
* ICD or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated eltroxine substituted myxoedema)
* Anemia (male: hemoglobin < 8.0; female: hemoglobin < 7.0 mmol/l)

Rapid-Heart:

Inclusion criteria - chronic hyperglycaemia cohort

* Informed and written consent
* Type 1 diabetes
* Age ≥18 years
* C-peptide negative (<0.2 nmol/l)
* Insulin treatment for ≥1 year
* HbA1C ≥63 mmol/mol

Inclusion criteria - well-controlled cohort

* Informed and written consent
* Type 1 diabetes
* Age ≥18 years
* C-peptide negative (<0.2nmol/l)
* Insulin treatment for ≥1 year
* HbA1C ≤53 mmol/mol

Exclusion criteria - both cohorts

* Arrhythmia diagnosed prior to or at the time of the screening visit
* ECG with left or right bundle branch block diagnosed prior to the screening visit.
* Implantable cardioverter defibrillator or pacemaker at the time of inclusion
* Heart failure diagnosed prior to the screening visit (left ventricular ejection fraction < 45%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated myxoedema)
* Anaemia (male: haemoglobin <8.0 mmol/l; female: haemoglobin <7.0 mmol/l)
* Treatment with anticoagulant or antiplatelet treatment
* Bleeding disorder diagnosed prior to the screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the global work during hypoglycemia in individuals with type 1 diabetes, type 2 diabetes, and without diabetes, respectively. | 255 minutes (Hypo-Heart 1) and 190 minutes (Hypo-Heart 2)
  Absolute change in the global work index measured by pressure-strain loop analysis during insulin-induced hypoglycemia compared to euglycemia in individuals with type 1 diabetes, type 2 diabetes, and without diabetes, respectively (Hypo-Heart 1 and Hypo-Heart 2).
  Study outcomes will be analyzed separately for each included study.

SECONDARY OUTCOMES:
Primary secondary outcome: Change in mechanical dyssynchrony during hypoglycemia in individuals with type 1 diabetes, type 2 diabetes, and without diabetes, respectively. | 255 minutes (Hypo-Heart 1) and 190 minutes (Hypo-Heart 2)
  Absolute change in mechanical dyssynchrony (defined as the standard deviation of regional time to peak strain) measured by speckle tracking echocardiography measured by pressure-strain loop analysis during insulin-induced hypoglycemia compared to euglycemia in individuals with type 1 diabetes, type 2 diabetes, and without diabetes, respectively (Hypo-Heart 1 and Hypo-Heart 2).
  Study outcomes will be analyzed separately for each included study.
Change in the global work during recovery in individuals with type 1 diabetes. | 255 minutes
  Absolute change in the global work index measured by pressure-strain loop analysis during recovery (post-hypoglycemic euglycemia and hyperglycemia) compared to euglycemia in individuals with type 1 diabetes (Hypo-Heart 1).
  Study outcomes will be analyzed separately for each included study.
Change in mechanical dyssynchrony during recovery in individuals with type 1 diabetes. | 255 minutes
  Absolute change in mechanical dyssynchrony (defined as the standard deviation of regional time to peak strain) measured by speckle tracking echocardiography measured by pressure-strain loop analysis during recovery (post-hypoglycemic euglycemia and hyperglycemia) compared to euglycemia in individuals with type 1 diabetes (Hypo-Heart 1).
  Study outcomes will be analyzed separately for each included study.
Change in the global work during hyperglycemia in individuals with type 1 diabetes, type 2 diabetes and without diabetes, respectively. | 255 minutes (Rapid Heart) and 190 minutes (Hypo-Heart 2)
  Absolute change in the global work index measured by pressure-strain loop analysis during hyperglycemia compared to euglycemia in individuals with type 1 diabetes, type 2 diabetes and without diabetes, respectively (Rapid Heart and Hypo-Heart 2).
  Study outcomes will be analyzed separately for each included study.
Change in mechanical dyssynchrony during hyperglycemia in individuals with type 1 diabetes, type 2 diabetes and without diabetes, respectively. | 255 minutes (Rapid Heart) and 190 minutes (Hypo-Heart 2)
  Absolute change in mechanical dyssynchrony (defined as the standard deviation of regional time to peak strain) measured by speckle tracking echocardiography measured by pressure-strain loop analysis during hyperglycemia compared to euglycemia in individuals with type 1 diabetes, type 2 diabetes and without diabetes, respectively (Rapid Heart and Hypo-Heart 2).
  Study outcomes will be analyzed separately for each included study.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, Principal Investigator — Steno Diabetes Center Copenhagen, Denmark
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark